CLINICAL TRIAL: NCT03935451
Title: A Randomized Controlled Trial on the Use of Postoperative Extended Venous Thromboprophylaxis in Patients With Inflammatory Bowel Disease: A Pilot Study
Brief Title: Postoperative Extended Venous Thromboprophylaxis in Inflammatory Bowel Disease
Acronym: EXPAND
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7043
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: IBD; Venous Thromboembolism; Crohn Disease; Ulcerative Colitis; Pulmonary Embolism; Colorectal Disorders
MeSH Terms: conditions — Venous Thromboembolism; Crohn Disease; Colitis, Ulcerative; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo group will receive a similarly appearing full supply of a twice daily placebo oral tablet.
  Interventions: Drug: Placebo Oral Tablet
- Experimental (Experimental): The treatment arm will receive a full supply of twice daily 2.5 milligram (mg) dosing of apixaban beginning on the first day of hospital discharge.
  Interventions: Drug: Apixaban 2.5 milligram

INTERVENTIONS:
Drug: Apixaban 2.5 milligram — 2.5 milligram daily dosing of Apixaban beginning on the first day of hospital discharge for a total of 30 days
  Arms: Experimental
Drug: Placebo Oral Tablet — placebo oral tablet that resembles the experimental drug. To be taken with the same frequency and duration
  Arms: Placebo

SUMMARY:
Inflammatory bowel disease (IBD) is a relatively common disease that effects all age groups and carries significant morbidity and mortality. The initial treatment typically involves both short and long term medication, however when this is not enough to adequately control the disease, surgery is often required. The high morbidity and mortality rates are in part due to the increased rates of venous thromboembolism (VTE) such as deep vein thrombosis (DVT) or pulmonary embolism (PE) which have been shown to develop more frequently in IBD patients compared to the general population. Undergoing abdominal surgery has also been shown to independently increase rates of DVT and PE and since the majority of patients with IBD will undergo surgery at least once in their lifetime, the relative increased risk of developing a VTE is very high. The majority of DVT and PE events in the postoperative IBD population will occur after discharge from hospital and therefore carries significant morbidity and mortality risk in a unmonitored setting. Several studies have demonstrated the benefits and safety of twice daily dosing of oral extended VTE prophylaxis agents in orthopedic and cancer postoperative patients following discharge from hospital. There have been no randomized studies which have evaluated the use of extended postoperative VTE prophylaxis in IBD patients. The purpose of this randomized placebo controlled pilot trial will be to evaluate the efficacy and safety of postoperative VTE prophylaxis in IBD patients following abdominal surgery. If this pilot trial demonstrates efficacy in reducing postoperative DVT and PE rates, safety and feasibility, clinicians will be armed with the knowledge to pursue a larger multicenter randomized trial with the intent of reducing overall morbidity and mortality in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Having documented pathological diagnosis of either Crohn's disease or ulcerative colitis.
* Open or laparoscopic abdominal gastrointestinal surgery
* Elective surgery
* Surgery occurring at Hamilton Health Sciences or St. Joseph's Healthcare Hamilton
* Negative urine beta-hCG for women of childbearing potential

Exclusion Criteria:

* Contraindication to use of postoperative thromboprophylaxis (ie. Previous bleeding on anticoagulation)
* Allergy to apixaban
* History of VTE
* Current clinically significant active bleeding, including GI bleeding
* Hepatic disease associated with coagulopathy and clinically relevant bleeding risk
* Severe renal impairment (eCrCl <30 ml/min), or undergoing dialysis
* Lesions or conditions at increased risk of clinically significant bleeding (e.g. recent GI bleeding, recent ischemic or hemorrhagic cerebral infarction, active ulcerative GI disease, recent brain, spinal or ophthalmological surgery, bronchiectasis or history of pulmonary bleeding, thrombocytopenia or functional platelet defects, congenital or acquired coagulation disorder)
* Receiving any of the following drugs:

  * Strong inhibitors of both CYP 3A4 and P-gp, such as azole-antimycotics (e.g. ketoconazole, itraconazole, voriconazole, or posaconazole), and HIV protease inhibitors (e.g. ritonavir)
  * Strong inducers of both CYP 3A4 and P-gp (e.g. rifampicin, phenytoin, carbamazepine, phenobarbital, or St. John's Wort)
  * Drug products affecting hemostasis (e.g. NSAIDs, ASA or other antiplatelet agents [e.g. ASA, clopidogrel, prasugrel, ticagrelor], SSRIs, or SNRIs)
  * Any other anticoagulant, including unfractionated heparin, LMWH, heparin derivatives, or oral anticoagulants (e.g. warfarin, dabigatran, rivaroxaban)
* Currently receiving therapy for any type of malignancy (e.g. colorectal, breast, lung)
* History of colorectal cancer
* Emergency surgery
* Patients with an indication for anticoagulation before surgery (atrial fibrillation, etc.)
* Enrolled in any other clinical trials or prospective studies where similar outcomes are measured
* Pregnant (i.e. positive pregnancy test and/or self-reported) and/or breastfeeding
* Women of childbearing potential unwilling/unable to participate in appropriate family planning during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post operative venous thromboembolism events (DVT/PE) in in patients with Inflammatory Bowel Disease | 3 months post operatively
  The primary efficacy outcome will be a composite of symptomatic proximal DVTs of the upper and lower extremities, splanchnic VTE, nonfatal PE (segmental or greater artery), and death from PE and death from any cause within 3 months following hospital discharge.
Incidence of bleeding while undergoing treatment with oral anticoagulant or placebo. | 3 months post operatively
  The primary safety outcome will be bleeding reported during treatment, including major bleeding, clinically relevant non-major (CRNM) bleeding, minor bleeding, and the composite of major bleeding and CRNM bleeding.

SECONDARY OUTCOMES:
Incidence of surgical complications related to post operative anticoagulation | 3 months post operatively
  The secondary outcome will include surgical complications related to anticoagulation (intra-abdominal bleeding, surgical site bleeding), and arterial thromboembolic events such as acute ischemic stroke, myocardial infarction, and other VTE (upper extremity and splanchnic veins).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
This study will not share any individual participant data with other researchers.